CLINICAL TRIAL: NCT07225153
Title: Goat Milk-Derived Formula Alternatives vs. Undiluted Goat Milk in Babies Unable to Exclusively Breastfeed: Analysis of Growth Metrics and Biological Markers
Brief Title: Goat Milk-Derived Formula vs. Undiluted Goat Milk in Infants Unable to Exclusively Breastfeed: Growth and Biomarker Analysis
Acronym: GMDFA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); University of Colorado, Boulder (Other); Baker Heart Research Institute (Other)
Responsible Party: Principal Investigator, Junaid Iqbal, Assistant Professor Research, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-11220-34303; D43TW007585 (NIH)
Record Dates: First submitted 2025-11-04; First posted 2025-11-05 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Malnutrition (Calorie); Infant Nutrition Disorder; Growth Flatering; Gut Microbiome; Lipidomics
Keywords: Infant nutrition; goat milk; Infant feeding practices; Breastfeeding; Breastfeeding Alternatives; Alternate feeding practices; Growth outcomes; Infant growth metrics; Gut microbiome; Gut inflammation biomarkers; Calprotectin; Lipocalin-2; Claudin-2; C-reactive protein (CRP); Randomized controlled trial; Rural Pakistan; Infant health; Malnutrition prevention; Lipidomics; Breast milk; Metagenomics
MeSH Terms: conditions — Malnutrition; Infant Nutrition Disorders; Breast Feeding

STUDY DESIGN:
Intervention Model Description: This is a three-arm, parallel-group, community-based randomized controlled trial designed to compare the effects of Goat Milk-Derived Formula Alternative (GMDFA), undiluted goat milk, and exclusive breastfeeding on infant growth, gut microbiome, and metabolic health. Infants will be randomly assigned to one of the three groups and followed concurrently for a 8-week intervention period. Each group will receive its assigned feeding regimen in parallel, with no crossover between groups.
Masking Description: This is an open-label trial due to the visible differences between feeding interventions (GMDFA, undiluted goat milk, and breastfeeding). Participants, caregivers, and field investigators will be aware of group assignments.
  However, to reduce potential bias, laboratory personnel conducting the microbiome, metagenomic, and lipidomic analyses will remain blinded to the feeding group assignments throughout sample processing and data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Goat Milk-Derived Formula Alternative (GMDFA) (Experimental): Infants in this arm will receive Goat Milk-Derived Formula Alternative (GMDFA) as their primary source of feeding for 08 weeks. Growth, safety, and biological markers will be assessed through anthropometric measurements and laboratory analyses, including microbiome, metagenomic, and lipidomic profiling.
  Interventions: Dietary Supplement: GMDFA
- Undiluted Goat Milk (Current Practice) (Active Comparator): Infants in this arm will receive undiluted goat milk according to local feeding practices, representing the current alternative to breastfeeding in the community. Growth and biological markers will be compared with the GMDFA and breastfed groups to evaluate safety and nutritional adequacy.
  Interventions: Other: Undiluted Goat Milk
- Breastfed Group (Reference Comparator) (No Intervention): Infants in this arm will be exclusively breastfed following WHO guidelines. No feeding intervention will be introduced. This group serves as the gold standard for comparison of growth metrics, microbiome composition, and metabolic biomarkers with the GMDFA and undiluted goat milk groups.

INTERVENTIONS:
Dietary Supplement: GMDFA — GMDFA (GOat Milk-Derived Formula Alternative) is a goat milk-based formulation designed as an affordable alternative to commercial infant formula. It is prepared by diluting goat's milk to a standardized protein and micronutrient concentration according to study protocol. Infants in this arm will receive GMDFA from enrollment (08-10 weeks) until 16-18 weeks of age under close monitoring for growth and safety outcomes.
  Arms: Goat Milk-Derived Formula Alternative (GMDFA)
Other: Undiluted Goat Milk — Infants will receive undiluted goat milk as per current local feeding practices for 8 weeks.
  Arms: Undiluted Goat Milk (Current Practice)

SUMMARY:
The goal of this clinical trial is to learn if Goat Milk-Derived Formula Alternatives (GMDFA) are safe and effective for infants who are unable to be exclusively breastfed. It will also study growth patterns, biological markers, and gut microbiome differences among infants receiving GMDFA, undiluted goat milk, or breast milk.

The main questions it aims to answer are:

1. Do infants receiving GMDFA show similar growth patterns to those who are breastfed?
2. Are biological markers of gut health and nutrition (such as calprotectin, lipocalin-2, CRP, and claudin) comparable between the groups?
3. How do feeding types (GMDFA, goat milk, or breast milk) influence the infant gut microbiome composition, metabolic pathways, and lipid profiles?
4. Is GMDFA a safe and nutritionally adequate feeding option for infants unable to be exclusively breastfed?

We will compare GMDFA, undiluted goat milk, and breast milk (reference group) to evaluate infant growth, gut health, and metabolic outcomes.

Participants will:

Be randomly assigned to one of three feeding groups: GMDFA, undiluted goat milk, or breastfed

Attend regular follow-up visits for growth measurements and sample collection (blood, stool, and breast milk where applicable)

Have feeding practices monitored and recorded through caregiver interviews and feeding logs

Additional Analyses:

Microbiome analysis: to identify gut bacterial diversity and composition across feeding groups Metagenomic analysis: to explore functional genes and metabolic pathways related to nutrition and gut health Lipidomic analysis: to assess differences in lipid and fatty acid profiles in breast milk, goat milk, and infant samples

DETAILED DESCRIPTION:
This community-based randomized controlled trial will evaluate the safety, nutritional adequacy, and biological effects of a Goat Milk-Derived Formula Alternative (GMDFA) among infants aged 8-10 weeks in Matiari, Pakistan, who are unable to exclusively breastfeed. The study includes three groups: (1) an intervention group receiving GMDFA prepared according to a standardized recipe developed for the study, (2) a control group receiving undiluted goat milk according to local feeding practices, and (3) an active comparator group of exclusively breastfed infants serving as a reference.

The intervention will last for 8 weeks. Primary and secondary outcomes will assess changes in lipidomic profiles, micronutrient status, gut inflammatory biomarkers (CRP, lipocalin-2, calprotectin, Claudin), and gut microbiome composition and diversity (Bifidobacterium, Firmicutes, Bacteroides, Clostridium, Lactobacillus). Anthropometric measurements including weight, length, and head circumference will be recorded at baseline and follow-up to evaluate infant growth outcomes.

The study aims to determine whether GMDFA provides a safe and nutritionally appropriate alternative to formula milk for infants who cannot be exclusively breastfed, with comparable biological and growth outcomes to breastfed infants. Findings from this study will inform the potential use of goat milk-based alternatives in low-resource settings where malnutrition and suboptimal breastfeeding rates are prevalent.

ELIGIBILITY:
Inclusion Criteria:

* • Infants aged = 08 -10 weeks with WAZ better than -1.8. (NIPS & ICF, 2019) Age Sex WAZ Weight in Kilograms 2 Month Boys WAZ>-1.8 4-5 kg 2 Month Girls WAZ>-1.8 4-5 kg Table 3: WAZ scores

  * Living in Matiari District.
  * Who has access to goat milk in their households.
  * The Breastfeeding group: Women who exclusively breastfeeding and not giving and sort of formula or animal derived milk.
  * Intervention Group: Women who do not breastfeed at all or give goat milk to their infants (2-3 feeds per day).
  * No birth deformities

Exclusion Criteria:

* • Infant birth weight < WAZ -1.8 i.e. weight-for-age based on established growth standards, such as the World Health Organization (WHO).

  * Birth deformities or disorders, such as genetic disorders, aerodigestive problems, or congenital anomalies.
  * Plan to migrate during the next six months.
  * We will exclude the women who exclusive breast feed and continue breast feeding for first 4 months.
  * If the child is enrolled or included in any other interventional trial.
  * Who does not have access to goat milk in their households.
  * Are medically disqualified: Any potential participant who is deemed medically unfit for enrollment, due to the presence of severe or unstable health conditions that could compromise safety or interfere with the study outcomes, will be excluded from participation

Ages: 8 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2025-08-30 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in lipidomic markers among infants receiving Goat Milk-Derived Formula Alternative (GMDFA) compared to undiluted goat milk and breastfeeding groups. | Baseline (enrollment) to 8 weeks after intervention
  To evaluate whether infants aged 8-10 weeks in Matiari who are unable to exclusively breastfeed and receive GMDFA show favorable changes in lipidomic profiles compared to those fed undiluted goat milk, and similar metabolic marker status compared to exclusively breastfed infants after 8 weeks of intervention.
Change in gut microbiome composition and diversity among infants receiving GMDFA compared to undiluted goat milk and breastfeeding groups. | Baseline (enrollment) to 8 weeks after intervention
  To determine whether infants aged 8-10 weeks in Matiari who are unable to exclusively breastfeed and receive Goat Milk-Derived Formula Alternative (GMDFA) exhibit distinct shifts in gut microbiome composition (Bifidobacterium, Firmicutes, Bacteroides, Clostridium, and Lactobacillus) and changes in alpha- and beta-diversity over 8 weeks, compared to those fed undiluted goat milk, and a microbiome profile similar to age-matched breastfed infants and healthy reference profiles from the same population.

SECONDARY OUTCOMES:
Infant growth measured by weight-for-age z-score (WAZ) | From baseline (enrollment) to 16-18 weeks of age
  Change in infant weight-for-age z-score from enrollment to 16-18 weeks of age, comparing GMDFA, breastfeeding, and undiluted goat milk groups.
Change in serum micronutrient levels among infants receiving GMDFA compared to undiluted goat milk and breastfeeding groups. | Baseline (enrollment) to 8 weeks after intervention
  To determine whether infants aged 8-10 weeks in Matiari who are unable to exclusively breastfeed and receive Goat Milk-Derived Formula Alternative (GMDFA) exhibit higher serum concentrations of essential micronutrients (vitamin A, vitamin B12, vitamin D, calcium, iron, and zinc) compared to those fed undiluted goat milk, and comparable micronutrient status to exclusively breastfed infants after 8 weeks of intervention.
Change in gut inflammatory biomarkers among infants receiving GMDFA compared to undiluted goat milk and breastfeeding groups. | Baseline (enrollment) to 8 weeks after intervention
  To assess whether infants aged 8-10 weeks in Matiari who are unable to exclusively breastfeed and receive Goat Milk-Derived Formula Alternative (GMDFA) show favorable changes in gut inflammatory markers (CRP, Lipocalin-2, Claudin, and Calprotectin) compared to those fed undiluted goat milk, and similar gut inflammatory marker status to exclusively breastfed infants after 8 weeks of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. junaid Iqbal, PhD, Principal Investigator — Aga Khan University; Syed Asad Ali, MPH, Study Director — Aga Khan University
Locations (1):
- MATIARI Research & Training Centre, Matiāri, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] George AD, Paul S, Wang T, Huynh K, Giles C, Mellett N, Duong T, Nguyen A, Geddes D, Mansell T, Saffery R, Vuillermin P, Ponsonby AL, Burgner D, Burugupalli S, Meikle PJ; Barwon Infant Study Investigator Team. Defining the lipid profiles of human milk, infant formula, and animal milk: implications for infant feeding. Front Nutr. 2023 Aug 30;10:1227340. doi: 10.3389/fnut.2023.1227340. eCollection 2023. PMID 37712002
- [Background] Vandenplas Y, Zolnowska M, Berni Canani R, Ludman S, Tengelyi Z, Moreno-Alvarez A, Goh AEN, Gosoniu ML, Kirwan BA, Tadi M, Heine RG, Cinnamon Study Investigator Group. Effects of an Extensively Hydrolyzed Formula Supplemented with Two Human Milk Oligosaccharides on Growth, Tolerability, Safety and Infection Risk in Infants with Cow's Milk Protein Allergy: A Randomized, Multi-Center Trial. Nutrients. 2022 Jan 26;14(3):530. doi: 10.3390/nu14030530. PMID 35276889
- [Background] Akter S, Nishu NA. Malnutrition among under-5 children and its determinants in the southwestern coastal region of Bangladesh: A community-based study. BMJ Open. 2025 Jan 14;15(1):e090174. doi: 10.1136/bmjopen-2024-090174. PMID 39809564
- [Background] Moreno-Avila IDM, Martinez-Linares JM, Garcia-Pintor S, Rubia-Ortega SM, Ortiz-Paneque J, El Messaoudi-Ouardani S, Cortes-Martin J. Perceptions on the Reasons Influencing the Choice and Abandonment of Exclusive Breastfeeding in Muslim and Christian Women: A Phenomenological Study. Nurs Health Sci. 2025 Sep;27(3):e70195. doi: 10.1111/nhs.70195. PMID 40695358
- [Background] Reinhardt K, Fanzo J. Addressing Chronic Malnutrition through Multi-Sectoral, Sustainable Approaches: A Review of the Causes and Consequences. Front Nutr. 2014 Aug 15;1:13. doi: 10.3389/fnut.2014.00013. eCollection 2014. PMID 25988116
- [Background] Omer S, Zakar R, Zakar MZ, Fischer F. The influence of social and cultural practices on maternal mortality: a qualitative study from South Punjab, Pakistan. Reprod Health. 2021 May 18;18(1):97. doi: 10.1186/s12978-021-01151-6. PMID 34006307
- [Background] Pietrzak-Fiecko R, Kamelska-Sadowska AM. The Comparison of Nutritional Value of Human Milk with Other Mammals' Milk. Nutrients. 2020 May 14;12(5):1404. doi: 10.3390/nu12051404. PMID 32422857
- [Background] Organization, W. H. (2005). Guiding principles for feeding non-breastfed children 6-24 months of age, World Health Organization.
- [Background] Organization, W. H. (2003). Complementary feeding: report of the global consultation, and summary of guiding principles for complementary feeding of the breastfed child, World Health Organization.
- [Background] Noh JW, Kim YM, Akram N, Yoo KB, Cheon J, Lee LJ, Kwon YD, Stekelenburg J. Factors Affecting Breastfeeding Practices in Sindh Province, Pakistan: A Secondary Analysis of Cross-Sectional Survey Data. Int J Environ Res Public Health. 2019 May 14;16(10):1689. doi: 10.3390/ijerph16101689. PMID 31091768
- [Background] Nayik GA, Jagdale YD, Gaikwad SA, Devkatte AN, Dar AH, Dezmirean DS, Bobis O, Ranjha MMAN, Ansari MJ, Hemeg HA, Alotaibi SS. Recent Insights Into Processing Approaches and Potential Health Benefits of Goat Milk and Its Products: A Review. Front Nutr. 2021 Dec 6;8:789117. doi: 10.3389/fnut.2021.789117. eCollection 2021. PMID 34938763
- [Background] Militao, E. M., Salvador, E. M., Silva, J. P., Uthman, O. A., Vinberg, S., & Macassa, G. (2022). Coping strategies for household food insecurity, and perceived health in an urban community in southern Mozambique: a qualitative study. Sustainability, 14(14), 8710.
- [Background] Kinsella HM, Hostnik LD, Toribio RE. Energy endocrine physiology, pathophysiology, and nutrition of the foal. J Am Vet Med Assoc. 2022 Oct 26;260(S3):S83-S93. doi: 10.2460/javma.22.08.0348. PMID 36288202
- [Background] Kandhro F, Kazi TG, Afridi HI, Baig JA, Lashari AA, Lashari A. Determination of toxic elemental levels in whey milk of different cattle and human using an innovative digestion method: risk assessment for children < 6.0 months to 5 years. Environ Sci Pollut Res Int. 2023 Mar;30(14):41923-41936. doi: 10.1007/s11356-022-25059-1. Epub 2023 Jan 14. PMID 36640239
- [Background] Kabir F, Iqbal J, Jamil Z, Iqbal NT, Mallawaarachchi I, Aziz F, Kalam A, Muneer S, Hotwani A, Ahmed S, Umrani F, Syed S, Sadiq K, Ma JZ, Moore SR, Ali A. Impact of enteropathogens on faltering growth in a resource-limited setting. Front Nutr. 2023 Jan 10;9:1081833. doi: 10.3389/fnut.2022.1081833. eCollection 2022. PMID 36704796
- [Background] Iqbal NT, Syed S, Sadiq K, Khan MN, Iqbal J, Ma JZ, Umrani F, Ahmed S, Maier EA, Denson LA, Haberman Y, McNeal MM, Setchell KDR, Zhao X, Qureshi S, Shen L, Moskaluk CA, Liu TC, Yilmaz O, Brown DE, Barratt MJ, Kung VL, Gordon JI, Moore SR, Ali SA. Study of Environmental Enteropathy and Malnutrition (SEEM) in Pakistan: protocols for biopsy based biomarker discovery and validation. BMC Pediatr. 2019 Jul 22;19(1):247. doi: 10.1186/s12887-019-1564-x. PMID 31331393
- [Background] Goraya MU, Li R, Mannan A, Gu L, Deng H, Wang G. Human circulating bacteria and dysbiosis in non-infectious diseases. Front Cell Infect Microbiol. 2022 Aug 24;12:932702. doi: 10.3389/fcimb.2022.932702. eCollection 2022. PMID 36093202
- [Background] Ahmed F, Malik NI, Zia S, Akbar AS, Li X, Shahid M, Tang K. Rural mothers' beliefs and practices about diagnosis, treatment, and management of children health problems: A qualitative study in marginalized Southern Pakistan. Front Public Health. 2023 Jan 4;10:1001668. doi: 10.3389/fpubh.2022.1001668. eCollection 2022. PMID 36684927
- [Background] Fantuz, F., et al. (2022). "Macro Minerals and Trace Elements in Milk of Dairy Buffaloes and Cows Reared in Mediterranean Areas." Beverages 8(3): 51.
- [Background] 8. Fantuz, F., et al. (2016). Macro-and micronutrients in non-cow milk and products and their impact on human health. Non-bovine milk and milk products, Elsevier: 209-261.
- [Background] Corden E, Siddiqui SH, Sharma Y, Raghib MF, Adorno W 3rd, Zulqarnain F, Ehsan L, Shrivastava A, Ahmed S, Umrani F, Rahman N, Ali R, Iqbal NT, Moore SR, Ali SA, Syed S. Distance from Healthcare Facilities Is Associated with Increased Morbidity of Acute Infection in Pediatric Patients in Matiari, Pakistan. Int J Environ Res Public Health. 2021 Nov 7;18(21):11691. doi: 10.3390/ijerph182111691. PMID 34770204
- [Background] 6. Borton, R. E. (2018). The Influence Of Social And Economic Factors On Breastfeeding And Rural Mothers, Illinois State University.
- [Background] Bhutta ZA, Berkley JA, Bandsma RHJ, Kerac M, Trehan I, Briend A. Severe childhood malnutrition. Nat Rev Dis Primers. 2017 Sep 21;3:17067. doi: 10.1038/nrdp.2017.67. PMID 28933421
- [Background] Bhutta ZA, Akseer N, Keats EC, Vaivada T, Baker S, Horton SE, Katz J, Menon P, Piwoz E, Shekar M, Victora C, Black R. How countries can reduce child stunting at scale: lessons from exemplar countries. Am J Clin Nutr. 2020 Sep 14;112(Suppl 2):894S-904S. doi: 10.1093/ajcn/nqaa153. PMID 32692800
- [Background] Arif S, Khan H, Aslam M, Farooq M. Factors influencing exclusive breastfeeding duration in Pakistan: a population-based cross-sectional study. BMC Public Health. 2021 Nov 3;21(1):1998. doi: 10.1186/s12889-021-12075-y. PMID 34732175
- [Background] Ali S, Ali SF, Imam AM, Ayub S, Billoo AG. Perception and practices of breastfeeding of infants 0-6 months in an urban and a semi-urban community in Pakistan: a cross-sectional study. J Pak Med Assoc. 2011 Jan;61(1):99-104. PMID 22368919
- [Background] Alliance for Maternal and Newborn Health Improvement (AMANHI) mortality study group. Population-based rates, timing, and causes of maternal deaths, stillbirths, and neonatal deaths in south Asia and sub-Saharan Africa: a multi-country prospective cohort study. Lancet Glob Health. 2018 Dec;6(12):e1297-e1308. doi: 10.1016/S2214-109X(18)30385-1. Epub 2018 Oct 22. PMID 30361107